CLINICAL TRIAL: NCT05119842
Title: Study on the Safety and Effectiveness of APrevent® VOIS Implants for Treatment in Patients With Unilateral Vocal Fold Paralysis (UVFP) - a Two-Part, Open-Label, Non-Randomized Multicenter Study
Brief Title: APrevent-VOIS-Implant-002 - a Two-Part, Open-Label, Non-Randomized Multicenter Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: APrevent Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APrevent-VOIS-Implant-002
Record Dates: First submitted 2021-11-04; First posted 2021-11-15 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Paralysis, Unilateral, Vocal Cord
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Intervention Model Description: The study will consist of two parts to assess safety, and effectiveness of the investigational device.
  Part A (Safety): In total 8 patients will be enrolled sequentially in three groups (N=1, N=2, N=5). An interval of at least 7 days between the groups will be left to allow the safety board to review individual patient's safety and demographic data. After completion of the first four patients and all three groups in Part A, an independent Data Safety Monitoring Board (DSMB) will recommend the initiation of study Part B based on the review of the safety data.
  Part B: In Part B of the study, the remaining 22 patients of the study will be enrolled non-sequentially.
  Part A and B (Effectiveness Population) will include: The part A patients will also be used for the confirmatory testing of the primary endpoint. At the end of the study safety of the investigational device will be assessed on patients of part A and B together.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Treatment with the VOIS Implant
  Interventions: Device: APrevent® VOIS-Implant

INTERVENTIONS:
Device: APrevent® VOIS-Implant — To compare the voice quality assessed by the change in G-Score from GRBAS-Scale between before and after permanent APrevent® VOIS implantation.

SUMMARY:
This is a prospective, 2-part, multi-center, open-label, non-randomized clinical trial to assess safety and effectiveness of APrevent® VOIS Implants for the treatment of patients with Unilateral Vocal Fold Paralysis (UVFP). In total 30 evaluable patients are planned to be enrolled.

DETAILED DESCRIPTION:
The APrevent® VOIS is intended to be permanently implanted during a type I thyroplasty in individuals suffering from permanent unilateral vocal fold paralysis of various etiologies. Four post-operative follow-up visits are planned: Week 1 (± 7 days), Week 7 (-7/+28 days), Month 6 (-14/+28 days) and Month 12 (-14/+28 days).

This 2-part study will consist of Part A to assess safety of the patients and the following Part B to assess the performance (effectiveness) of the investigational device. In Part A of the study 8 patients will be enrolled sequentially within three groups (N=1, N=2, N=5). After enrolment and 1st Follow-up Visit of each group, a Local Safety Board will review safety and study data. No preliminary/interim analysis of safety and effectiveness data will be performed before the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 80 years
* Diagnosed with permanent UVFP and insufficient glottal closure
* A significant voice disorder as measured by perceptual rating (Grade ≥2 GRBAS Scale) and Voice Handicap Index (VHI-30 score >33)
* Ability to comprehend the full nature and purpose of the study, including possible risks and side effects
* Ability to co-operate with the Investigator and to comply with the requirements of the entire study
* Availability to volunteer for the entire study duration, willing to adhere to all protocol requirements and willing and able to give informed consent for participation

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the clinical investigation may influence the result of the clinical investigation, or the participant's ability to participate in the clinical investigation
* Scheduled elective surgery or other procedures requiring general anaesthesia during clinical investigation
* Bilateral vocal fold paralysis
* Had injection medialization laryngoplasty with the injectable still being within the double length of the maximum resorption time frame as stated in their approval or as supported by literature.
* Presence of structural vocal fold lesions such as polyp or nodules
* Presence of oropharyngeal or laryngeal tumors
* Patients with diagnosed severe obstructive sleep apnea (OSA)
* Status post total cordectomy
* Previous laryngeal framework surgery (any type of thyroplasty, arytenoid adduction)
* Status post tracheostomy
* Presence of acute systemic infection at time of screening or shortly before surgery
* Significant non-laryngeal speech abnormality (severe dysarthria determined by a panel of trained speech therapists)
* Severe coagulopathy
* Females who are pregnant, lactating or planning pregnancy are excluded from the investigation
* Patients with bil. Gr. III-IV hypertrophic tonsils
* Diabetes mellitus with poor control and poor wound healing history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in G-Score from GRBAS-Scale | 7weeks
  Change in G-Score from GRBAS-Scale from before to 7 weeks after permanent APrevent® VOIS implantation

SECONDARY OUTCOMES:
Change in Maximum Phonation Time (MPT, unit seconds) from before to 7 weeks after permanent APrevent® VOIS implantation. | 7 weeks
  MPT will be measured in seconds using a digital stop clock. The patient will be asked to say a prolonged vowel "a" for as long as possible after maximal inspiration. The best out of three trials in seconds will be chosen for comparison.

OTHER OUTCOMES:
R-Score from GRBAS-Scale from before to 7 weeks after permanent APrevent® VOIS implantation. | 7 weeks
  R-Score from GRBAS-Scale from before to 7 weeks after permanent APrevent® VOIS implantation.
B-Score from GRBAS-Scale (range [0…3]) from before to 7 weeks after permanent APrevent® VOIS implantation | 7 weeks
  B-Score from GRBAS-Scale from before to 7 weeks after permanent APrevent® VOIS implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Leonhard, Dr, Principal Investigator — Study principal investigator
Locations (7):
- United States (4):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Medical University of Vienna, Vienna, Austria
- Germany (2):
  - SRH Wald-Klinikum Gera, Gera
  - University Medical Center, Hamburg

IPD SHARING:
Plan to Share IPD: No